# Informed Consent Form Cover Page for ClinicalTrials.Gov Record

Official Study Title: Impact of combined medication and behavioral treatment in young children with comorbid ASD and ADHD

NCT #: NCT03242772

Duke University Health System (DUHS) Protocol #: Pro00085179

Document Version Date (DUHS IRB Reference Date of Consent Form): 24-APR-2021

Document Name/Consent Type: Minor Main Study consent



A+ Treatment

Duke Center for Autism Research Program

## **Concise Summary**

The purpose of this research study (A+ Treatment) is to determine whether a combined therapy (an investigational stimulant drug and a behavioral intervention based on parent coaching designed for children with Autism Spectrum Disorder (ASD) can improve behavioral and developmental functioning of children with Attention Deficit Hyperactivity Disorder (ADHD) and ASD more than a placebo and the same behavioral intervention for ASD. The parent coaching intervention is based on a model called "Early Start Denver Model" (ESDM) which involves strategies that can be used during daily activities to promote social interaction, language, and behavioral regulation (e.g. reduce tantrums). Participants will first complete screening and a behavioral assessment that includes a blood draw, physical exam, collection of medical and behavioral information, questionnaires, and activities measuring attention, brain activity, and social interaction.

If eligible for the study, children will be assigned by a computer (that doesn't consider any personal information about them) to receive either the investigational medication or placebo, both which are in tablet form, dissolve in the mouth, and are called "study drug" in the rest of this form. The entire study is about 3 months with an optional follow-up remote questionnaire assessment. After receiving a diagnostic and cognitive assessment and medical/behavioral assessment visit (about 3 weeks), for the next 8 weeks, your child will receive either behavioral intervention plus the medication or behavioral intervention plus placebo. During the 10 weeks of treatment, your doctor will adjust your child's medication if needed and regularly assess any side effects. The behavioral intervention will be weekly 1-hour sessions of ESDM-based parent coaching. A week after completing the behavioral intervention, your child will participate in another behavioral assessment, described in more detail below. There are optional follow-up parent questionnaires that can be completed remotely at 24 weeks.

Possible risks include potential side effects from the active drug including common side effects such as loss of appetite, trouble sleeping, stomach pain, nausea, vomiting, nervousness and fever and very rare side effects including fast or irregular heartbeat, prolonged erections, seizures or hallucinations.

Potential benefits: Your child may benefit by receiving diagnostic and cognitive evaluations that are conducted as part of this study. Your family could also benefit from the ESDM-based parent coaching. The study drug may or may not reduce some of your child's ADHD symptoms. It is more likely that the active study drug will reduce ADHD symptoms than the placebo study drug.

If you are interested in learning more about this study, please continue to read below.


#### INTRODUCTION

You and your child are being asked to take part in this research study because your child is enrolled in the Duke Autism Center of Excellence ("Duke ACE Center") research program and you have expressed interest participating in the A+ Treatment study for children with ASD and ADHD.

DUHS RB
IRB NUMBER: Pro00085179
IRB REFERENCE DATE: 04/24/2021
IRB EXPIRATION DATE: 04/04/2022



A+ Treatment

Duke Center for Autism Research Program

Please read this consent form carefully and take your time making a decision. The nature of the study, including the risks and benefits, are explained below. Please ask the staff member who provided this consent form to explain any words or information that you do not clearly understand.

Participation in a research study is always completely voluntary. If you do agree to have your child participate, you can change your mind and may withdraw your child from the study at any time. Any services that your child receives through a Duke University-affiliated (or non-Duke affiliated) clinic or primary care provider will not be affected by your decision about your child's participation in this study. We encourage you to talk with your family and friends before you and your child decide to take part in this research study. Please tell the study doctor or study staff if your child is taking part in another research study.

This part of the Duke ACE Center program is called the "A+ Treatment Study" and it is overseen by Dr. Lauren Franz, the study's Principal Investigator, and Dr. Tara Chandrasekhar, the study's physician. The A+ Treatment Project and the Duke ACE Center are sponsored by a grant from the National Institutes of Health (NIH). Portions of Dr. Franz's and Dr. Chandrasekhar's and their research team's salaries are by this grant.

## WHO WILL BE MY CHILD'S DOCTOR ON THIS STUDY?

If you and your child decide to participate, Dr. Franz, Dr. Chandrasekhar, or one of the other study doctors will be your child's study doctor and may be in contact with your child's regular health care provider (if you choose) throughout the time that you and your child are in the study and afterwards, if needed.

## WHY IS THIS STUDY BEING DONE?

Approximately half of children with ASD also have ADHD. We are studying whether the combination of parent-coaching behavioral intervention and a stimulant drug that helps children focus (Adzenys®XR-ODT) can improve ASD and ADHD symptoms for young children with both ADHD and ASD more than behavioral intervention alone.

Adzenys®XR-ODT has been approved by the U.S. Food and Drug Administration (FDA) to help children with ADHD alone in patients ages 6 and above. It has not yet been studied in children younger than 6 years old. The Adzenys®XR-ODT is identical to another stimulant drug, Adderall, which has been approved by the FDA for children without specifying age and has been used for many years. The goal of this study is to help doctors in the future better treat children with both ASD and ADHD.

## **HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?**

Approximately 48 children and their parent(s) will take part in this study at Duke.

DUHS RB
IRB NUMBER: Pro00085179
IRB REFERENCE DATE: 04/24/2021
IRB EXPIRATION DATE: 04/04/2022

| Parent/Guardian | Initials |
|-----------------|----------|



A+ Treatment

Duke Center for Autism Research Program

## WHAT IS INVOLVED IN THE STUDY?

If you agree for you and your child to be in this study, you will be asked to sign and date this consent form.

The Duke A+ Treatment study will evaluate your child's health, social and language abilities, brain activity, and how they interact with you and play. There will be 12 in-person visits to our clinic. The visits and study activities are described below. At 24 weeks, you will have the option to fill out some questionnaires about your child's behavior remotely (you do not need to come to the university).

Visits will include diagnostic and cognitive assessments to determine preliminary eligibility for A+ Treatment as well as a health screener to see if you and your child can participate in our study. The health screener will be its own separate visit outlined below.

#### **Health Screener**

You and your child will be asked to come to the clinic and a doctor will decide if your child is eligible for the treatment part of the study. This visit will take around 4-6 hours.

- The doctor will collect some medical and behavioral information about your family and your child and problems your child may be having.
- o We will measure your child's heart rate, blood pressure, weight, height and temperature.
- We will measure the electrical activity in your child's heart to make sure your child's heart is healthy. This test is called an Electrocardiography (ECG) and it will record the electrical activity of your child's heart through small electrode patches that a research staff member will attach to the skin of his/her chest, arms, and/or legs.

After this visit and the cognitive and diagnostic assessments, if the study doctor decides that your child can be in the study and you wish to participate; you and your child will be enrolled into the study.

#### Visits 4 - 12

At the next visit your child will be assigned by a computer that does not consider any personal information about your child to receive either placebo or Adzenys®XR-ODT (extended release orally-disintegrated tablet) for 10 weeks. A placebo is an inactive substance given in the same form as the active study drug. The placebo tablet will look and taste exactly the same as the active medication. These tablets are placed on your child's tongue and will melt within 1-2 minutes. Slightly more kids will be assigned to receive the study drug with the active medication than with the placebo. Your child will have approximately a 54% chance of receiving the study drug. Neither you nor the study doctor will know what your child receives. However, in the event of an emergency, your child's study doctor will have the ability to find out which group your child is in if he/she feels that knowing that information will affect your child's care during the emergency. In the rest of this consent form both placebo and active study drug


DUHS |RB IRB NUMBER: Pro00085179 IRB REFERENCE DATE: 04/24/2021 IRB EXPIRATION DATE: 04/04/2022





A+ Treatment

Duke Center for Autism Research Program

(Adzenys®XR-ODT) will be called the "study drug". Once the study drug treatment period is complete, one of our unblinded study team members will contact you to tell you if your child was on the medication or placebo so you can better make decisions about continuation of care for your child.

Approximately 2 weeks later, you will begin 8 weekly 1- hour sessions of ESDM Informed Parent Coaching. During these visits, the doctor and research staff will meet with you to monitor the drug and any side effects. A week (Visit 12) after completing the ESDM Informed Parent Coaching sessions, your child will be assessed again using the same assessments that were completed at baseline, including collection of medical and behavioral information, questionnaires, and activities measuring attention, brain activity, and social interaction.

# **Study Drug Monitoring**

During the first several weeks after receiving medication, the study doctor will start at a low dose of study drug (Adzenys®XR-ODT or placebo-ODT) and slowly increase the dose until the best dose is reached for your child. You and your child will be coming to the clinic or receiving phone calls and/or emails by the study doctor and/or study staff to make sure your child is not having any problems with the study drug during this time. If you or your child feels the study drug is causing problems or is not helpful at any time, you are not obligated to continue to take the study drug. You and your child also have the option of continuing the behavioral intervention and assessment visits, even though you stop the study medication. Or you and your child can stop the study completely.

## To monitor how your child is doing on the study drug, the following things will occur:

- The research staff will monitor your child's heart rate, blood pressure, height and weight.
- The study doctor and or study staff will ask you and your child about any possible benefits or bad effects or other problems that your child may have experienced while taking the drug.
- The study doctor will perform a physical exam to identify any potential side effects from the study medication.
- You will be asked to rate your child's attention in a number of different areas to help the study doctor determine the potential benefits of the study medication.

Then the study doctor will talk to you about options related to your child's dose of the study drug, trying to find the dose that results in the most improvement of ADHD symptoms and the fewest side effects. We hope that we will be able to identify the best dose of study medication 2-3 weeks after dispensing the study drug.

Parent-Delivered Early Start Denver Model (P-ESDM) - Informed Coaching

DUHS |RB IRB NUMBER: Pro00085179 IRB REFERENCE DATE: 04/24/2021 IRB EXPIRATION DATE: 04/04/2022

 Parent/Guardian Initials\_\_\_\_\_





A+ Treatment

Duke Center for Autism Research Program

A therapist trained in parent coaching of ESDM will meet with you and your child 8 times, once a week, for about 60 minutes to coach you in the use of strategies to promote social and language abilities and behavioral regulation (e.g. reduce tantrums). Another family member may also attend these sessions, but it is important that you come to each therapy visit. This is to ensure that you learn how all the different ESDM Informed Parent Coaching strategies work together and so that the therapist and you can work together to learn which strategies work best for you and to try to make strategies that are more challenging easier to use.

ESDM Informed Parent Coaching is a therapy developed from an evidence-based form of behavioral therapy called ESDM that uses principles of Applied Behavior Analysis (ABA) to promote language, social interaction, and behavioral regulation. During each coaching session, the therapist will check in with how things are going with your child, briefly talk about the strategies to be learned and practiced during that coaching session, and then give you feedback as you work with your child trying the strategy and other techniques. Finally, towards the end of the appointment, you and the therapist will talk about specific things to try during the next week.

#### **Assessment Visits**

You and your child will complete several questionnaires and activities to help us understand how your child is progressing in paying attention to things going on around him/her, social and language skills, and behavior. These physician visits will take around 3-4 hours. These activities are described below. They will be repeated 1 week after completing 8 weeks of ESDM Informed Parent Coaching. It is important that you, not some other caretaker, complete these forms and come to these visits so that we can see and measure the changes in your child over time as accurately as possible.

## • Questionnaires and Interviews

- Prior to starting treatment and after completing behavioral therapy, you will be asked to complete a set of questionnaires (sent electronically or completed in person), which include questions about your child's social skills, language, emotional expression, interests, and other behaviors, such as sleep habits.
   Some of these will also ask how you and your child are feeling and doing, and about your experiences in the study.
- There will also be parent interviews where we will ask you about the behaviors that you observe your child doing regularly in your home where we can't observe your child ourselves.

## Assessment of social interaction, communication, and attention

 Your child will participate in activities that involve playing with toys and observing how he/she responds to the examiner. Some of these activities will be audio- and video-taped so we can be sure each examiner is interacting in the same way as the other examiners.

DUHS |RB IRB NUMBER: Pro00085179 IRB REFERENCE DATE: 04/24/2021 IRB EXPIRATION DATE: 04/04/2022

| Parent/Guardian | Initials |
|-----------------|----------|



A+ Treatment

Duke Center for Autism Research Program

- Other assessments of social interaction and communication. We will audio- and video-tape most of these interactions so we can go back and count how often specific behaviors occur to get more precise measurements that might show change over time
  - We will observe and videotape how your child naturally plays with you and a specific set of toys.
  - We will measure how you and your child moves about in the room using a video tracking camera, called EthoVision® XT.
  - We will measure where your child is looking while he/she is watching movies shown on a special computer monitor. The camera that records where your child is looking is called Tobii TX300.
  - You and your child may view a set of short engaging videos on an iPhone or tablet, and the camera on the iPhone or tablet will record your child's facial expressions and responses to the videos.

## Brain activity

Before treatment begins and one week after completing behavioral intervention, , we will measure your child's brain activity using EEG recordings to see if and how your child's brain activity changes when watching either pictures of faces or pictures of objects. A net made of a set of wet sponges will be placed on your child's head while your child watches a TV screen that will show short videos with pictures and sounds, each video lasting about 5 minutes with breaks between each video.

At 24 weeks, you will have the option of completing additional questionnaires about your child's behavior remotely either through a phone call or e-mail (at home).

The study doctor may determine that additional visits, procedures or tests are clinically necessary even though they are not specifically listed as part of the study in order to be sure your child is receiving the best possible medical care. You can refuse the study doctor's recommendations for these things, but refusal may affect you and your child's participation in the study and could result in you and your child being taken out of the study.

#### **Future Contact**

If you enroll your child in the Duke ACE program you may receive the following information occasionally:

- Information cards via email (or mail, with pre-stamped envelope) to inform us of any changes in your contact information (address, e-mail address, and/or phone number),
- Newsletters to update you on ongoing activities of the Duke ACE Center,


- Holiday and birthday cards,
- Invitations to special community events hosted by the Center (such as sports clinics and artwork contests),

DUHS |RB IRB NUMBER: Pro00085179 IRB REFERENCE DATE: 04/24/2021 IRB EXPIRATION DATE: 04/04/2022



A+ Treatment

Duke Center for Autism Research Program

 Information about other research-related opportunities, including the Registry for Autism Research.

# **Contact with the A+ Treatment Study Team**

The study will use email (acetreatment@duke.edu) to communicate with you about visit scheduling and follow-ups as needed. Because using your personal e-mail does not provide a completely secure and confidential means of communication, please do not use it if you wish to keep your communication private. Instead, let us know and we will communicate with you only through the telephone or Duke MyChart. You may also call the study physician, Dr. Tara Chandrasekhar at (919)-627-1652.

# Video and Audio Recording Activities

Audio and video recordings of assessments of you and your child (e.g., in behavioral, play-based activities, or interviews conducted with you and/or your child) will be used for data analysis, and quality monitoring.

If you agree, these videotapes may also be used for training and/or educational purposes. Please indicate your choice by writing your initials next to your selection below (this will not affect the participation of you and your child in the study).

| Yes, I agree to allow my and my child's videotaped session to be used for training purposes. |
|---|
| Yes, I agree to allow my and my child's videotaped session to be used for educational purposes. |
| OR |
| No, I do not agree to allow my and my child's videotaped session to be used for training and/or educational purposes. |

#### **HOW LONG WILL I BE IN THIS STUDY?**

Total participation is expected to require 12 weeks plus an optional remote visit with questionnaires at 24 weeks.

## WHAT ARE THE RISKS OF THE STUDY?

#### Risks of Active Study Drug

As a result of your participation in this study, your child may be at risk for the following sideeffects from the active study drug. You should discuss these with the study doctor and, if you

DUHS RB
IRB NUMBER: Pro00085179
IRB REFERENCE DATE: 04/24/2021
IRB EXPIRATION DATE: 04/04/2022



A+ Treatment

Duke Center for Autism Research Program

want, with your child's regular health care provider. Adzenys®XR-ODT may cause some, all or none of the side-effects listed below.

#### More common

- Loss of appetite
- Trouble sleeping
- Weight loss
- Abdominal pain
- Nausea
- Vomiting
- Nervousness
- Fever

## Less Likely

- Irregular heartbeat
- Other heart-related problems like high blood pressure
- Seizures
- Hair loss
- Blurred vision
- Tics
- Hallucinations
- Prolonged erections

## **Controlled Drug**

- A. Adzenys®XR-ODT is under Schedule II in the FDA's list of controlled substances. This means that:The drug or other substances have a high potential for abuse
- B. The drug or other substances have currently accepted medical use in treatment in the United States, or currently accepted medical use with severe restrictions
- C. Abuse of the drug or other substances may lead to severe psychological or physical dependence

Therefore, for you and your child's safety we ask that under no circumstances that this drug be given to anyone else, including yourself. We will be closely monitoring the number of tablets we give you for your child at each visit and the number of tablets returned to our clinic at each medication visit, to be sure your child is taking the medication as directed. If you have any issues over the course of the study, please do not hesitate to contact either the study coordinators, Dr. Franz at (919) 681-0023, or the study physician, Dr. Chandrasekhar at (919)-627-1652.

For more information on the FDA's list of controlled substances please follow the link provided:

DUHS RB
IRB NUMBER: Pro00085179
IRB REFERENCE DATE: 04/24/2021
IRB EXPIRATION DATE: 04/04/2022

 Parent/Guardian Initials\_\_\_\_\_





A+ Treatment

Duke Center for Autism Research Program

https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfcfr/CFRSearch.cfm?CFRPart=1308.

## **Risks of Placebo**

There is a possibility that the study drug and/or placebo won't reduce your child's ADHD symptoms and/or won't help your child respond better to ESDM Informed Parent Coaching. This possibility may be greater with the placebo study drug than the active study drug, but this has not been tested/seen in young children with both ADHD and ASD. There is also the possibility that if your child weren't in the study and took a different medication or treatment for ADHD symptoms that your child would respond better to that medication or have fewer side effects with that medication or treatment than with the study drug. Currently there are no medications that are proven to improve the fundamental challenges with social communication and repetitive behaviors in ASD. This is why we encourage you to work with a doctor outside the study if you want to look into other treatments for ADHD or ASD after week 24 of the study.

## **Risk of Discontinuing Prior Medication**

Any ADHD medication in the form of stimulants, or atomoxetine, must be discontinued prior to starting the study medication. Of course, discontinuing any prescribed medication entails some risk. There is a possibility that there will be an increase in ADHD symptoms. If these symptoms become intolerable at any point, please do not hesitate to contact us, as consent for study is an ongoing process. Dr. Franz or the study physician will be available to discuss with you whether the potential benefits of being in the trial (outlined below) outweigh the benefits of restarting your child's prior medication or obtaining other community based behavioral treatments. If you still feel restarting medication will be the best option for your child, you can withdraw from the study knowing that this does not keep your child from receiving other services from Duke outside of the study.

## **Other Medicine**

- The study physician may prescribe melatonin (6mg/night) if your child is still having trouble sleeping even with a reduction in dose of the study medication and if you want to do this. Melatonin is a hormone that your body produces naturally to help control sleep/wake cycles. Melatonin is sometimes taken as a dietary supplement in a pill or readily dissolvable form to help people with trouble sleeping. Although studies with melatonin have shown no serious adverse effects, there are a few possible side effects:
  - o Melatonin can make symptoms of depression worse
  - Melatonin can raise blood pressure in people who are taking other medications
  - Using melatonin might increase the risk of having a seizure


 If melatonin doesn't help your child sleep better and you want to try a different medication to help with sleep, the study physician may prescribe either a drug called clonidine or one called diphenhydramine, also known as Benadryl. Clonidine is a

DUHS |RB IRB NUMBER: Pro00085179 IRB REFERENCE DATE: 04/24/2021 IRB EXPIRATION DATE: 04/04/2022

| Parent/Guardian | Initials |
|-----------------|----------|
|-----------------|----------|



A+ Treatment

Duke Center for Autism Research Program

medicine that can be used for high blood pressure or during the day for ADHD. However, it tends to cause sleepiness, so many doctors use it to help children sleep. Clonidine can have the following side effects

- Drowsiness
- o Dizziness
- o Tiredness
- Irritability
- Light headedness
- Lower heart rate
- Lower blood pressure
- High blood pressure if suddenly discontinue clonidine
- Diphenhydramine is an antihistamine used to relieve allergy and cold symptoms. It is also shown to help people relax and fall asleep. Common side effects of diphenhydramine include:
  - Drowsiness
  - Dizziness
  - Constipation
  - Upset stomach
  - Blurred vision
  - Dry mouth
- Clonazepam is an anti-anxiety medication. Common side effects of clonazepam include:
  - Drowsiness
  - Poor coordination
  - Unsteadiness while walking
  - Depression

If your child is prescribed melatonin, clonidine, clonazepam or diphenhydramine, it will not be provided for or paid by the study.

## **Drug and Food Interactions**

For your child's safety, you must tell the study doctor about all the prescribed medical foods and drugs, herbal products, over-the-counter (OTC) drugs, vitamins, natural remedies, and alcohol that your child is taking before you start the study and before starting to take any of these products while you are on the study.

We will watch over your child closely by checking your child's vital signs at each visit. We will initially check your child's heart activity and ensure it is healthy. At visits we will also be

DUHS RB
IRB NUMBER: Pro00085179
IRB REFERENCE DATE: 04/24/2021
IRB EXPIRATION DATE: 04/04/2022

 Pare



A+ Treatment

Duke Center for Autism Research Program

monitoring any problems with the study drug your child may have and perform regular physical exams.

## Risks of Electrocardiogram (ECG)

Possible side effects of the ECG are skin irritation, itching, and redness from the ECG electrode pads. Let the study coordinator or physician know of any previous skin conditions or discomfort your child might have before the pads are applied.

## **Other Risks**

There is a possibility that you or your child may become frustrated during study tasks. We will try to make the tasks and task directions as easy as possible. Your child can take as many breaks as he/she needs during assessments. Some of the questions we will ask you or your child as part of this study may make you or your child feel uncomfortable. You or your child may refuse to answer any of the questions and you or your child may take a break at any time during the study. You or your child may stop your participation in this study at any time.

There is also the potential risk of loss of confidentiality. Every effort will be made to keep your information confidential; however, this cannot be guaranteed.

## Risks related to your child's ASD and ADHD

Your child may experience a worsening of symptoms that may be because of their condition alone, or because they are not taking their regular medicine, or because of a lot of other factors that may not be related to this study. This may be more likely if your child is taking the placebo study drug rather than the active study drug. The study doctor will try to minimize these risks by carefully monitoring your child during the study. In cases of severe worsening of symptoms that place your child or those around him/her at risk, your child may require inpatient hospitalization. If the study doctor feels that your child is at serious risk for hurting him/herself or others, he/she can ask a judge to allow your child to be hospitalized against your and/or your child's will.

There may be risks, discomforts, drug interactions or side effects that are not yet known.

#### ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

If you and your child agree to take part in this study, your child may benefit by receiving some of the diagnostic and cognitive evaluations that are conducted as part of this study. Your family could also benefit from the ESDM informed parent coaching and learning how to use strategies for promoting social skills, language, and behavioral regulation.

It is also possible that the study medication may help improve some of your child's ADHD symptoms. However, we will not be providing the study drug after the last in-person visit, the study doctor will discuss whether you want to continue to pursue ADHD treatment for your


DUHS RB
IRB NUMBER: Pro00085179
IRB REFERENCE DATE: 04/24/2021
IRB EXPIRATION DATE: 04/04/2022



A+ Treatment

Duke Center for Autism Research Program

child. If you do, we will be happy to provide a referral to a medical provider not associated with the study.

There are still potential benefits if your child is in the placebo group. Your child will still be receiving a parent-coaching behavioral therapy along with other behavioral assessments as previously mentioned. If at any point you feel that restarting prior ADHD medication will be more beneficial to your child than continuing participation in the study drug treatment portion of the study, we hope you will continue to participate in the remaining efficacy assessments in the trial. We will stop providing the study drug to your child if you choose to pursue other medication treatments for ADHD for your child outside the study, but will continue to provide parent coaching if you agree to participate in ongoing efficacy and safety assessments.

Finally, we also hope that in the future the information learned from this study will benefit other people with both ASD and ADHD.

#### WHAT ALTERNATIVES ARE THERE TO PARTICIPATION IN THIS STUDY?

Instead of being in this study, you and your child have the following alternatives:

- Other early intervention therapy for ASD
- Other medication or behavior therapy for ADHD in young children
- Have your child try medicine for associated symptoms, such as anxiety or irritability

Please talk to your child's doctor about these and perhaps other options.

## WILL MY CHILD'S INFORMATION BE KEPT CONFIDENTIAL?

Participation in research involves some loss of privacy. This study will collect information that might directly identify you and your child, such as names, dates of birth, addresses and health related information. We understand that information about you and your child's health is personal, and we are committed to protecting the privacy of that information. We will do our best to make sure that information about you and your child is kept confidential, but we cannot guarantee total confidentiality. You and your child's personal information may be viewed by individuals involved in this research and may be seen by people including those collaborating, funding, and regulating the study. Collaborators include individuals who are not part of Duke University. We will share only the minimum information in order to conduct the research. You and your child's personal information may also be given out if required by U.S. or State law. Examples of information that we are legally required to disclose include abuse or neglect of a child.

As part of the study, results of your child's study-related data and procedures may be reported to the NIH and its affiliates. In addition, your child's records may be reviewed in order to meet federal or state regulations. Reviewers may include representatives from the Food and Drug Administration (FDA), representatives and affiliates of the NIH, and the Duke University Health


DUHS RB
IRB NUMBER: Pro00085179
IRB REFERENCE DATE: 04/24/2021
IRB EXPIRATION DATE: 04/04/2022



A+ Treatment

Duke Center for Autism Research Program

System Institutional Review board, and others as appropriate. If any of these groups review your child's research record, they may need to review your child's entire medical records.

The Duke ACE Center will use a third-party web-based application called Q-Global from Pearson, Inc. to collect data and score the responses for one of the questionnaires in this study. To properly score this assessment, only your child's date of birth and his/her study ID will be entered along with your responses. The minimal amount of information will be submitted over a secure (industry-standard Secure Socket Layer (SSL)) Internet connection to Q-Global for purposes of accurately scoring the questionnaire. The information provided to Q-Global is subject to its terms of use. The Q-Global web-based platform is secure (data is encrypted using industry-standard SSL technology and compliant with established HIPAA Security Regulations as well as changes to HITECH Act effective March 2013 which applies to Business Associates to health care providers). However, as with any website platform or software, there may be potential security risks and Duke cannot guarantee that the website is free of risk.

Except when required by law, and as otherwise explained in this consent document, you or your child will not be identified by name, address, telephone number, or any other direct personal identifier in records disclosed outside of Duke University Health System (DUHS). All data can only be accessed by a secure password which will be locked away by authorized personnel. The database will be stored on a secure server at the Duke School of Medicine. Study team members are required to log in with a unique username and password to access the study database. Before being granted access to the study database, staff complete training on protecting confidentiality and sign confidentiality agreements. The database will include all the information that we collect during the course of the study and it will also include information such as your child's date of birth, gender, and date of each study visit. It also will contain your child's name and contact information in a dashboard. All hard copies of your child's records will be kept in locked file cabinets. Only people who need access to your child's data to do their job will have access to it. Any paper records will be stored in locked office.

This project is part of a larger set of projects that are part of the Duke Autism Center of Excellence funded by the National Institute of Child Health and Human Development. Data collected by this study will be shared with investigators who are part of the Duke Autism Center of Excellence. This will allow us to learn more by combining data across different projects that are part of the Duke Autism Center of Excellence program.

Some information collected about your child in this research study will be used only for the study and will be kept in a research study record separate from your child's medical record. Some research information may also be part of your child's medical record. You and your child will only have access to information about whether your child received the placebo or the study drug during the randomized double-blind portion of the study after all participants have

DUHS |RB IRB NUMBER: Pro00085179 IRB REFERENCE DATE: 04/24/2021 IRB EXPIRATION DATE: 04/04/2022

 Parent/Guardian Initials\_\_\_\_\_



A+ Treatment

Duke Center for Autism Research Program

completed the research study and the main study results have been analyzed. Some research information such as test results and psychological assessment reports will be available to your physicians if needed for your child's care.

The study results will be retained in your child's research record for six years after the study is completed or until your child reaches the age of 21, whichever is longer. At that time either the research information not already in your child's medical record will be destroyed or information identifying your child will be removed from such study results at DUHS. Any research information in your child's medical record will be kept indefinitely.

This information may be further disclosed by NIMH (National Institute of Mental Health), the funding agency of this study. If disclosed by the funding agency, the information is no longer covered by federal privacy regulations. If this information is disclosed to outside reviewers for audit purposes, it may be further disclosed by them and may not be covered by federal privacy regulations. NIMH is a part of the NIH.

While the information and data resulting from this study may be presented at scientific meetings or published in a scientific journal, your and your child's name or other personal information will not be revealed.

Some people or groups who receive your and your child's health information might not have to follow the same privacy rules. Once your and your child's information is shared outside of Duke, we cannot guarantee that it will remain private. If you decide to share your or your child's private information with anyone not involved in the study, the federal law designed to protect your and your child's health information privacy may no longer apply to the information you have shared. Other laws may or may not protect sharing of private health information.

#### **NDAR**

Data from this study may be submitted to the National Data for Autism Research (NDAR). NDAR is a data repository run by the NIMH that allows researchers studying children's health to collect and share de-identified information with each other. A data repository is a large database where information from many studies is stored and managed. De-identified information means that all personal information (such as name, address, and phone number) is removed and replaced with a code number. With an easier way to share, researchers hope to learn new and important things about children's health more quickly than before.

During and after the study, we will send de-identified information to NDAR. Other researchers nationwide can then file an application with the NIMH to obtain access to your or your child's de-identified study data for research purposes. Experts at the NIMH who know how to protect health and science information will look at every request carefully to minimize risks to your privacy.

DUHS RB
IRB NUMBER: Pro00085179
IRB REFERENCE DATE: 04/24/2021
IRB EXPIRATION DATE: 04/04/2022

 Parent/Guardian Initials\_\_\_\_\_





A+ Treatment

Duke Center for Autism Research Program

You may not benefit directly from allowing your information to be shared with NDAR. The information provided to NDAR may help researchers around the world treat future children and adults with mental illnesses so that they have better outcomes. NIMH will also report to Congress and on its web site about the different studies that researchers are conducting using NDAR data. However, you will not be contacted directly about the data you contributed to NDAR.

You may decide now or later that you do not want to share your or your child's information using NDAR. If so, contact Dr. Franz and she or a research study staff member will tell NDAR, which can stop sharing the research information. However, NDAR cannot take back information that was shared before you changed your mind. If you would like more information about NDAR, this is available on-line at http://data-archive.nimh.gov.

#### **Duke Patient**

As part of this study, your child will become a Duke patient. Dr. Franz and her study team will ask your child to have certain tests. Some of these tests and/or procedures would have been done as part of your child's regular care. She will use these test results both to treat your child and to complete this research. These test results will be recorded in your child's medical record and will be reported to the research team and representatives and affiliates of the funding agency. Some results of tests and studies done solely for this research study and not as part of your child's regular care will be included in your child's medical record.

#### **Other Disclosures**

A pediatric cardiologist (heart doctor) will review your child's ECG to determine if there might be possible concerns about your child's heart beat based on your child's age. When we collect your child's blood for general blood safety assessments, we will send the blood to an external laboratory called Laboratory Corporation of America Holdings, more commonly known as Labcorp. Labcorp will also need access to your child's date of birth in order to ensure that the results they report are accurate.

Neither the pediatric cardiologist nor Labcorp will receive any identifying information other than your child's date of birth. They will not have your child's name, medical record number or any other information.

## **Certificate of Confidentiality**

The Department of Health and Human Services (HHS) has issued a Certificate of Confidentiality to further protect your privacy. With this Certificate, the investigators may not disclose research information that may identify you in any Federal, State, or local civil, criminal, administrative, legislative, or other proceedings, unless you have consented for this use.

DUHS RB
IRB NUMBER: Pro00085179
IRB REFERENCE DATE: 04/24/2021
IRB EXPIRATION DATE: 04/04/2022




A+ Treatment

Duke Center for Autism Research Program

Research information protected by this Certificate cannot be disclosed to anyone else who is not connected with the research unless:

- 1) There is a law that requires disclosure (such as to report child abuse or communicable diseases but not for legal proceedings);
- 2) You have consented to the disclosure, including for your medical treatment; or
- 3) The research information is used for other scientific research, as allowed by federal regulations protecting research subjects.

Disclosure is required, however, for audit or program evaluation requested by the agency that is funding this project or for information that is required by the FDA.

You should understand that a Confidentiality Certificate does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it. This means that you and your family must also actively protect your own privacy.

Finally, you should understand that the investigator is not prevented from taking steps, including reporting to authorities, to prevent serious harm to yourself or others.

## WHAT ARE THE COSTS TO YOU?

There will be no additional costs to you or your child as a result of being in this study. However, routine medical care for your child's condition (care your child would have received whether or not your child was in this study) will be charged to you or your insurance company. You may wish to contact your insurance company to discuss this further. If anti-anxiety medication is requested by the parent/caregiver for the child's blood draw, you will need to pick this up before the visit at your pharmacy after our study doctor has prescribed it. In order to make sure that tests and studies done solely for research purposes are charged correctly, we will carefully monitor your Duke Hospital and Clinic charges as long as you are participating in this study. These tests and studies are not a part of routine care, and people who are not part of the study do not usually have them performed. Please ask Dr. Chandrasekhar or another study doctor if you would like to know more about which tests and studies are being done solely for research purposes.

The study drug will be provided free of charge for your child's use in this study up until week 10. At the conclusion of the first phase of the study (week 10), or if you or your child decide to withdraw from the study, you must return all unused study drug to Dr. Chandrasekhar or

DUHS RB
IRB NUMBER: Pro00085179
IRB REFERENCE DATE: 04/24/2021
IRB EXPIRATION DATE: 04/04/2022

 Parent/Guardian Initials\_\_\_\_\_



A+ Treatment

Duke Center for Autism Research Program

another study doctor. Dr. Chandrasekhar or another study doctor may request that you and your child return to complete the tests that would ordinarily occur when a person completes the study. If you decide at the end of the 10-week period/end of study that you wish to continue using the drug or put your child on the study drug, we will be happy to provide a referral to a another care physician not associated with the study. We will not be providing the ADHD drug nor will we provide any more coaching after study completion.

#### WHAT ABOUT COMPENSATION?

You and your child will be compensated up to a total of \$600 for participating in this study. You will be reimbursed \$50 for each of the 12 visits (health screener, physician visits, and ESDM Informed Parent Coaching visits). Participants will be compensated (\$50) for the optional follow-up questionnaires at week 24. Transportation costs ( within a 2 hour driving distance 1-way) can also be provided on a case by case basis, to reliably get to study visits if necessary.

Payment received as compensation for participation in research is considered taxable income to the research subject. If payment to an individual totals \$600 or more in any one calendar year, Duke University is required to report this information to the Internal Revenue Service (IRS). Research subject payments to a non-employee of Duke University adding up to \$600 or more during any calendar year will result in a 1099 (Miscellaneous Income) form being issued to the individual and a copy sent to the IRS.

## WHAT ABOUT RESEARCH RELATED INJURIES?

Immediate necessary medical care is available at Duke University Medical Center in the event that your child is injured as a result of your child's participation in this research study. However, there is no commitment by Duke University, Duke University Health System, Inc., or your Duke physicians to provide monetary compensation or free medical care to you in the event of a study-related injury.

For questions about the study or research-related injury, contact Dr. Franz at (919) 681-0023 or Dr. Chandrasekhar at (919)-681-0018 during regular business hours and (919)-627-1652 for Dr. Chandrasekhar after hours and on weekends and holidays.

# WHAT ABOUT MY RIGHTS TO DECLINE PARTICIPATION OR WITHDRAW FROM THE STUDY?

You and your child may choose not to be in the study, or, if you and your child agree to be in the study, you or your child may withdraw from the study at any time. If you or your child withdraw from the study, no new data about your child will be collected for study purposes other than data needed to keep track of your child's withdrawal, unless the data concern an adverse event related to the study. If such an adverse event occurs, we may need to review your child's entire medical record. All data that have already been collected for study purposes, and any new information about an adverse event related to the study, will be

DUHS |RB IRB NUMBER: Pro00085179 IRB REFERENCE DATE: 04/24/2021 IRB EXPIRATION DATE: 04/04/2022

 Parent/Guardian Initials\_\_\_\_\_



A+ Treatment

Duke Center for Autism Research Program

included in the research database. All data that have already been collected will be kept solely for study purposes and will be sent to the study sponsor.

You or your child's decision not to participate or to withdraw from the study will not involve any penalty or loss of benefits to which you and your child are entitled, and will not affect your child's access to health care at Duke. Signing this consent form is not a condition for receiving any medical care outside the study. However, if you or your child decides to stop participating in the study, we encourage you to talk to your child's doctor first. If you do decide to withdraw, we ask that you contact Dr. Franz in writing and let her know that you are withdrawing from the study. Her email address is: <a href="mailto:lauren.franz@duke.edu">lauren.franz@duke.edu</a> and her phone number is (919) 681-0023.

If you use email please be aware that you may be at potential risk for a loss of confidentiality because email is not a secure means of communication.

In addition, you must return all unused study drug to the study physician, Dr. Chandrasekhar, or her staff. She may also ask you and your child to complete the tests that would ordinarily occur when a person completes the study.

Your child's study doctor may decide to discontinue your child's participation in this study if your child's condition gets worse, if your child has serious side effects, or if your child's study doctor determines that it is no longer in your child's best interest to continue. The funding agency or regulatory agencies may stop this study at any time without your or your child's consent. Reasons why this might occur include because your child has had an unexpected reaction, or has failed to follow instructions, or because the entire study has been stopped. If this occurs, you will be notified and your child's study doctor will discuss other options with you.

If you do not sign this consent form and your child is a Duke patient, your child will continue to receive care from your healthcare provider, but not as a part of this study.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify your child. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

For questions about the study or a research-related injury, or if you have problems, concerns, questions or suggestions about the research, Dr. Franz at (919) 681-0023 or (919)-627-1652 for Dr. Chandrasekhar (another doctor on the study) after hours and on weekends and holidays.

DUHS RB
IRB NUMBER: Pro00085179
IRB REFERENCE DATE: 04/24/2021
IRB EXPIRATION DATE: 04/04/2022

 Parent/Guardian Initials\_\_\_\_\_

Form M0345



# Consent to Participate in a Research Study

A+ Treatment

Duke Center for Autism Research Program

For questions about your or your child's rights as a research participant, or to discuss problems, concerns or suggestions related to the research, or to obtain information or offer input about the research, contact the Duke University Health System Institutional Review Board (IRB) Office at (919) 668-5111.

#### STATEMENT OF CONSENT

"The purpose of this study, procedures to be followed, risks and benefits have been explained to me. I have been allowed to ask the questions I have, and my questions have been answered to my satisfaction. I have been told whom to contact if I have additional questions. I have read this consent form and agree to participate and allow my child to be in this study with the understanding that I may withdraw him/her or myself at any time. We have discussed the study with my child, who agrees to be in the study. I have been told that I will be given either a paper signed copy of this consent form or an electronic version, which will be sent to the email address (es) I choose to include below."

| Signature of Parent/Guardian #1 | Date | Time |
|-------------------------------------------------|------|----------|
| Name of Parent/Guardian #1 | | |
| Signature of Parent/Guardian #2 (if applicable) | Date | Time |
| Name of Parent/Guardian #2 (if applicable) | | |
| Signature of Person Obtaining Consent | Date | <br>Time |
| Name of Person Obtaining Consent | | |